CLINICAL TRIAL: NCT06364592
Title: Effect of Electroacupuncture for Dysmenorrhea Secondary to Adenomyosis: an Exploratory Pilot Study
Brief Title: Electroacupuncture for Dysmenorrhea Secondary to Adenomyosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Liu Zhishun, Chief Physician, Dean of Acupuncture Department, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-011-KY
Record Dates: First submitted 2024-04-02; First posted 2024-04-15 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Dysmenorrhea; Adenomyosis; Electroacupuncture
Keywords: Dysmenorrhea; Adenomyosis; Electroacupuncture
MeSH Terms: conditions — Dysmenorrhea; Adenomyosis | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Electroacupuncture, Then Sham Electroacupuncture (Experimental): Fifteen participants will first receive electroacupuncture for two consecutive menstrual cycles. After a washout period of one menstrual cycle, they then will receive sham electroacupuncture for another two consecutive menstrual cycles.
  Interventions: Device: Electroacupuncture; Device: Sham Electroacupuncture
- Sham Electroacupuncture, Then Electroacupuncture (Sham Comparator): Fifteen participants will receive sham electroacupuncture for two consecutive menstrual cycles. After a washout period of one menstrual cycle, they then will receive electroacupuncture for another two consecutive menstrual cycles.
  Interventions: Device: Electroacupuncture; Device: Sham Electroacupuncture

INTERVENTIONS:
Device: Electroacupuncture — Hwato brand disposable acupuncture needles (size 0.30 × 40 mm and 0.30 × 75 mm) and SDZ-V electroacupuncture apparatus will be used. Acupoints of Ciliao (BL32), Shiqizhui (EX-B8), and Sanyinjiao (SP6) will be used for participants.
  The needles will be inserted to 60-70mm in BL32 and 25-30mm in EX-B8 and SP6. Needle manipulation will be conducted (except for BL32) to achieve deqi sensation. Then paired electrodes from the electroacupuncture apparatus will be attached transversely to the needle handles at bilateral BL32 and SP6. The electroacupuncture stimulation will last for 30 minutes with a continuous wave of 5Hz and a current intensity of 1 to 5mA. Current intensity was adjusted according to the patients' individual tolerance.Treatment will start within one week before the onset of menstruation and stop before the end of menstruation, three sessions per menstrual cycle in total (ideally every two to three days and at least one session during menstruation period).
Device: Sham Electroacupuncture — Hwato brand disposable acupuncture needles (size 0.25 × 40 mm and 0.30 × 25 mm) and SDZ-V electroacupuncture apparatus will be used. Sham acupoints of BL32, EX-B8 and SP6 will be used for every participants.
  The needles will be inserted to 2-3mm in sham acupoints. Procedures, electrode placements, and other treatment settings were the same as in the electroacupuncture group but with no electricity output or needle manipulation for de qi.

SUMMARY:
The aim of this study is to preliminarily evaluate the is to assess the effects and safety of electroacupuncture for moderate to severe dysmenorrhea secondary to adenomyosis.

ELIGIBILITY:
Inclusion Criteria:

* Meeting the diagnosis criteria of dysmenorrhea secondary to adenomyosis.
* Female patients aged between 18 and 50.
* Dysmenorrhea lasting for 3 consecutive menstrual cycles or more.
* At least three consecutive menstrual cycles with an interval of 24 to 38 days, differing by less than 7 days, and menstrual periods lasting 2 to 8 days before screening.
* At least 2 days of worst pain score ≥4 on Numerical Rating Scale during the screening period.
* Having not used medications, other than rescue medicine, or therapies for dysmenorrhea secondary to adenomyosis for at least 1 month before randomization, and consenting not to use throughout the process of the research.
* Volunteering to participate the trial and signing written informed consent.

Exclusion Criteria:

* Diagnosed with Endometriosis or having a history of endometriosis-related surgery
* Currently taking hormonal medications, including: a.use of GnRH agonists within 6 months before the screening period; b. use of progestins or danazol and other long-acting hormones within 3 months before the screening period; c. use of oral contraceptive-like short-acting hormones within one month before the screening period;
* Having clinically significant gynecologic condition such as clinically significant endometrial pathology, persistent complex ovarian cyst larger than 3 cm or simple ovarian cyst larger than 5 cm, or single fibroid 4 cm or larger or more than 4 fibroids measuring at least 2 cm or symptomatic submucosal fibroid of any size.
* having an IUD.
* HB < 90G/L.
* Having any other chronic pain syndrome that required chronic analgesic or other chronic therapy.
* Having a current history of undiagnosed abnormal genital bleeding.
* Malignant tumors (including the reproductive system and other systems).
* Combined with severe diseases in the cardiac, respiratory, renal, liver, and hematopoietic systems, psychiatric disorder and/or cognitive disorders.
* Pregnant, breast feeding, planning a pregnancy within the next 7 months.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-21 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The change from baseline in the numerical rating scale (NRS) score on the worst pain | The menstruation period of Cycle 1, Cycle 2, Cycle 3, Cycle 4, Cycle 5 and Cycle 6 (each cycle is 24-38 days)]
  Participants will rate their worst pain during menstruation period of each menstrual cycle on a 0-10 NRS scale, where 0 refers to no pain and 10 refers to the worst pain imaginable. The highest worst pain score of the each cycle will be taken as final NRS score on the worst pain.

SECONDARY OUTCOMES:
The change from baseline in the numerical rating scale (NRS) score on the average pain | The menstruation period of Cycle 1, Cycle 2, Cycle 3, Cycle 4, Cycle 5, Cycle 6 and Cycle 7 (each cycle is 24-38 days)]
  Participants will rate their average pain during menstruation period of each menstrual cycle on a 0-10 NRS scale, where 0 refers to no pain and 10 refers to the worst pain imaginable. The final NRS score on average pain is defined as the mean of the average pain scores of each cycle.
The change from baseline in the numerical rating scale (NRS) score on the worst pain. | The menstruation period of Cycle 1, Cycle 4 and Cycle 7 (each cycle is 24-38 days)]
  Participants will rate their worst pain during menstruation period of each menstrual cycle on a 0-10 NRS scale, where 0 refers to no pain and 10 refers to the worst pain imaginable. The highest worst pain score of the each cycle will be taken as final NRS score on the worst pain.
Proportion of participants with at least 30% reduction of numerical rating scale (NRS) score on average pain. | The menstruation period of Cycle 1, Cycle 2, Cycle 3, Cycle 4, Cycle 5, Cycle 6 and Cycle 7 (each cycle is 24-38 days)]
  Participants will rate their average pain during menstruation period of each menstrual cycle on a 0-10 NRS scale, where 0 refers to no pain and 10 refers to the worst pain imaginable. The final NRS score on average pain is defined as the mean of the average pain scores of each cycle.
Proportion of participants with at least 30% reduction of numerical rating scale (NRS) score on the worst pain. | The menstruation period of Cycle 1, Cycle 2, Cycle 3, Cycle 4, Cycle 5, Cycle 6 and Cycle 7 (each cycle is 24-38 days)]
  Participants will rate their worst pain during menstruation period of each menstrual cycle on a 0-10 NRS scale, where 0 refers to no pain and 10 refers to the worst pain imaginable. The highest worst pain score of the each cycle will be taken as final NRS score on the worst pain.
The change from baseline in the Pictorial Blood Loss Assessment Chart (PBAC) score. | The menstruation period of Cycle 1, Cycle 2, Cycle 3, Cycle 4, Cycle 5, Cycle 6 and Cycle 7 (each cycle is 24-38 days)]
  After using each piece of sanitary napkin from the beginning to the end of each menstrual period, participants record it in a diary card according to the Pictorial Blood Loss Assessment Chart (PBAC) score. To ensure accuracy, participants are instructed to use sanitary napkins of the same size. The PBAC includes two parts of scoring records: the size of blood stain area in a sanitary napkin and lost blood clots.
The change from baseline in the the Cox Menstrual Symptom Scale (CMSS). | The menstruation period of Cycle 1, Cycle 2, Cycle 3, Cycle 4, Cycle 5, Cycle 6 and Cycle 7 (each cycle is 24-38 days)]
  The Cox Menstrual Symptom Scale (CMSS) consists of 18 items related to dysmenorrhea symptoms, such as lower abdominal pain, nausea, and headache, and each item is scored on a 5-point scale to measure severity and duration. Higher score corresponds to more severe dysmenorrhea symptoms.
The change from baseline in the Short Form Endometriosis Health Profile Questionnaire (EHP-5). | The last week of Cycle 1, Cycle 2, Cycle 3, Cycle 4, Cycle 5, Cycle 6 and Cycle 7 (each cycle is 24-38 days)]
  The Short Form Endometriosis Health Profile Questionnaire (EHP-5) is also commonly used to assess quality of life in patients with adenomyosis. The Questionnaire consists of 12 questions answered by a score of 1-5 points, the higher the score, the lower the quality of life.
The change from baseline in the total and sub scores of Hospital Anxiety and Depression Scale (HADS). | The last week of Cycle 1, Cycle 2, Cycle 3, Cycle 4, Cycle 5, Cycle 6 and Cycle 7 (each cycle is 24-38 days)]
  Hospital Anxiety and Depression Scale (HADS) consists of 14 items, divided into two 7 item subscales to reeect a state of generalized anxiety and the depression. The respondent rates each item on a 4-point scale ranging from 0 (absence) to 3 (extreme presence).

OTHER OUTCOMES:
Proportion of participants with positive expectance assessment | Before the first treatment session of electroacupuncture and sham electroacupuncture.
  Participants will be asked what do you think the condition of dysmenorrhea will be in two menstrual cycles?
Blinding assessment | Within 5 minutes after the last treatment in Cycle 3 and Cycle 6 (each cycle is 24-38 days).
  Participants will be ask "do you think you have received traditional electroacupuncture in the past two cycles?"
Adherence assessment | The menstruation period of Cycle 2, Cycle 3, Cycle 5 and Cycle 6 (each cycle is 24-38 days).
  Adherence will be assessment via counting treatment sessions. Those complete over 80% treatment sessions will be defined as of good adherence.
The change from baseline in the dose of rescue medicine. | The menstruation period of Cycle 1, Cycle 2, Cycle 3, Cycle 4, Cycle 5, Cycle 6 and Cycle 7 (each cycle is 24-38 days)]
  The dose of rescue medicine that participants use to relieve dysmenorrhea-related pain.

CONTACTS AND LOCATIONS:
Overall Officials: Zhishun Liu, Principal Investigator — Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Locations (1):
- Guang'anmen Hospital, China Academy of Chinese Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data and data dictionary will be available with the publication until six months after publication.
  A formal request should be sent to zhishunjournal@163.com with a methodologically sound proposal.
  Researchers whose proposal has been approved will sign a data access agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be available with the publication until six months after publication.
Access Criteria: A formal request should be sent to zhishunjournal@163.com with a methodologically sound proposal. Researchers whose proposal has been approved.
  Researchers whose proposal has been approved will sign a data access agreement.